CLINICAL TRIAL: NCT06091254
Title: A Phase 3, Open-label, Randomized Study to Compare the Efficacy and Safety of Odronextamab (REGN1979), an Anti-CD20 X Anti-CD3 Bispecific Antibody Versus Investigator's Choice in Previously Untreated Participants With Follicular Lymphoma (OLYMPIA-1)
Brief Title: A Trial to Learn if Odronextamab is Safe and Well-Tolerated and How Well it Works Compared to Rituximab Combined With Different Types of Chemotherapy for Adult Participants With Follicular Lymphoma
Acronym: OLYMPIA-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1979-HM-2298; 2022-502660-20-00 (EU CTIS Number)
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Follicular Lymphoma (FL)
Keywords: Non-Hodgkin lymphomas (NHLs); Indolent NHL; B-cells NHL (B-NHL); Follicular lymphoma; Odronextamab
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Prednisolone; Methylprednisolone; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Odronextamab (Experimental): Part 1 is a safety run-in. All participants will receive odronextamab.
  In part 2 participants will be randomly assigned in a 1:1 ratio to receive odronextamab followed by odronextamab maintenance.
  Interventions: Drug: Odronextamab
- Rituximab + Investigator's Choice Chemotherapy (Active Comparator): Part 2 only, participants will be randomized 1:1 to receive rituximab in combination with chemotherapy followed by rituximab maintenance.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone/prednisolone; Drug: Bendamustine

INTERVENTIONS:
Drug: Odronextamab — Administered by intravenous infusion (IV)
  Other Names: REGN1979
  Arms: Odronextamab
Drug: Rituximab — Rituximab will be administered by IV, or subcutaneously (SC)
  Other Names: Rituxan
  Arms: Rituximab + Investigator's Choice Chemotherapy
Drug: Cyclophosphamide — Administered by IV as part of Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (CHOP) chemotherapy, or Cyclophosphamide, Vincristine, Prednisone (CVP) chemotherapy
  Other Names: Cytoxan
  Arms: Rituximab + Investigator's Choice Chemotherapy
Drug: Doxorubicin — Administered by IV as part of CHOP chemotherapy
  Other Names: Adriamycin
  Arms: Rituximab + Investigator's Choice Chemotherapy
Drug: Vincristine — Administered by IV as part of CHOP, and CVP chemotherapy
  Other Names: Oncovin
  Arms: Rituximab + Investigator's Choice Chemotherapy
Drug: Prednisone/prednisolone — Administered orally (PO) as part of CVP chemotherapy
  Other Names: Deltasone/Omnipred
  Arms: Rituximab + Investigator's Choice Chemotherapy
Drug: Bendamustine — Administered by IV as part of chemotherapy (Rituximab-Bendamustine)
  Other Names: Treanda
  Arms: Rituximab + Investigator's Choice Chemotherapy

SUMMARY:
This study is researching an experimental drug called odronextamab, referred to as study drug. The study is focused on participants with previously untreated follicular lymphoma (a type of non-Hodgkin lymphoma or NHL).

This study will be made up of two parts: Part 1 (non-randomized) and Part 2 (randomized - controlled).

The aim of Part 1 of the study is to see how safe and tolerable the study drug is when given alone.

The aim of Part 2 of the study is to see how the study drug works compared to rituximab (called the "comparator drug") and chemotherapy (the current standard of care for NHL). Standard of care means the usual medication expected and used when receiving treatment for a condition.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)
* How the study drug affects quality of life and ability to complete routine daily activities.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of Cluster of Differentiation 20^+ (CD20^+) FL Grade 1-3a, stage II bulky or stage III / IV
2. Need for treatment as described in the protocol
3. Have measurable disease on cross-sectional imaging documented by diagnostic imaging Computed Tomography (CT) or Magnetic Resonance Imaging (MRI)
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
5. Adequate bone marrow function and hepatic function, as described in the protocol

Key Exclusion Criteria:

1. Central Nervous System (CNS) lymphoma or leptomeningeal lymphoma
2. Histological evidence of transformation to a high-grade or diffuse large B-cell lymphoma
3. Waldenström Macroglobulinemia (WM, lymphoplasmacytic lymphoma), Grade 3b follicular lymphoma, chronic lymphocytic leukemia, or small lymphocytic lymphoma
4. Treatment with any systemic anti-lymphoma therapy
5. Infections and allergy/hypersensitivity to study drug or excipient, as described in the protocol

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2028-02-19 (Estimated); Study Completion 2031-11-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) for odronextamab | Up to 35 days
  Part 1
Incidence of Treatment-Emergent Adverse Events (TEAEs) of odronextamab | Up to 2 years
  Part 1
Severity of TEAEs of odronextamab | Up to 2 years
  Part 1
Complete Response at 30 months (CR30) as assessed by independent central review | Up to 30 months
  Part 2

SECONDARY OUTCOMES:
Concentrations of odronextamab in serum | Up to 30 months
  Part 1
Incidence of Anti-Drug Antibodies (ADAs) to odronextamab over the study duration | Up to 30 months
  Part 1
Magnitude of ADAs to odronextamab over the study duration | Up to 30 months
  Part 1
Objective response as assessed by the investigator | Up to 30 months
  Part 1
Progression-Free Survival (PFS) as assessed by independent central review | Up to 5 years
  Part 2
Event-Free Survival (EFS) as assessed by independent central review | Up to 5 years
  Part 2
Overall Survival (OS) | Up to 5 years
  Part 2
Overall mean change in physical function [European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire 30 (EORTC-QLQ-C30)] | Up to 5 years
  Part 2 The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a global health status (GHS)/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
CR30 as assessed by local investigator | Up to 30 months
  Part 2
PFS as assessed by the local investigator | Up to 5 years
  Part 2
EFS as assessed by the local investigator | Up to 5 years
  Part 2
Objective response assessed by local investigator | Up to 30 months
  Part 2
Objective response assessed by independent central review | Up to 30 months
  Part 2
Duration Of Response (DOR) assessed by independent central review | Up to 5 years
  Part 2
DOR assessed by local investigator | Up to 5 years
  Part 2
Time To Next anti-lymphoma Treatment (TTNT) | Up to 5 years
  Part 2
Incidence of TEAEs | Up to 2 years
  Part 2
Severity of TEAEs | Up to 2 years
  Part 2
Odronextamab concentrations in serum during the induction period | Up to 30 months
  Part 2
Odronextamab concentrations in serum during the maintenance period | Up to 30 months
  Part 2
Incidence of ADAs to odronextamab over the study duration | Up to 30 months
  Part 2
Magnitude of ADAs to odronextamab over the study duration | Up to 30 months
  Part 2
Overall mean changes in scores of patient reported outcomes (PROs), as measured by the validated instruments EORTCQLQ- C30 | Up to 5 years
  Part 2 The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a global health status (GHS)/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
Overall mean changes in scores of PROs, as measured by the validated instruments Functional Assessment of Cancer Therapy-Lymphoma (FACT-LymS) | Up to 5 years
  Part 2 The FACT-Lym lymphoma subscale (LymS) includes 15 items to assess NHL-related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). Higher scores are associated with a worse quality of life.
Overall mean changes in scores of PROs, as measured by the validated instruments EuroQol-5 Dimension-5 Level Scale (EQ-5D- 5L) | Up to 5 years
  Part 2 The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: "no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems". The EQ VAS records the participant's self-rated health on a vertical visual analogue scale where the endpoints are labeled "Best imaginable health state" and "Worst imaginable health state".
Change in Patient Global Impression of Severity (PGIS) | Up to 5 years
  Part 2 The PGIS includes a single-item to assess how a patient perceives the overall severity of cancer symptoms over the past 7 days. Patients will choose the response that best describes the severity of their overall cancer symptoms with options on a 5-point scale ranging from 1 (No symptoms) to 4 (Very Severe).
Change in Patient Global Impression of Change (PGIC) | Up to 5 years
  Part 2 The PGIC item includes a single-item to assess how a patient perceives their overall change in health status since the start of study treatment. Patients will choose from response options on a 7-point scale ranging from 1 (Much Better) to 7 (Much worse); 1- Much Better, 2-Moderately Better, 3-A Little Better, 4-About the Same, 5-A Little Worse, 6-Moderately Worse, 7-Much Worse.
Change in score of the GP5 item in the participant population | Up to 5 years
  Part 2 A single item Global Population item 5 (GP5) of the validated FACT-G questionnaire will be used to assess from the participant perspective the overall impact of treatment side-effect. The question item is on a 5-point scale ranging from "not at all" (0) to "very much" (4).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (187):
- United States (20):
  - University of Arizona Cancer Center, Tucson, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UC Irvine Health, Orange, California
  - Investigative Clinical Research of Indiana, Noblesville, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Icahn School of Medicine at Mt Sinai, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Clinical Research Alliance Inc, Westbury, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Center for Oncology and Blood Disorders, Houston, Texas
  - HOPE Cancer Center of East Texas, Tyler, Texas
  - Huntsman Cancer Institute - Oncology Division, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Prohealth Care Inc, Waukesha, Wisconsin
- Australia (7):
  - Ingham Institute, Liverpool, New South Wales
  - Icon Cancer Centre - Wesley, Auchenflower, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Health, Clayton, Victoria
  - Epworth Freemasons, East Melbourne, Victoria
  - St Vincent's Hospital - Melbourne, Fitzroy, Victoria
  - Alfred Hospital and Monash University, Melbourne, Victoria
- Austria (5):
  - Ordensklinikum Linz, Linz, Osterreich
  - Ordensklinikum Linz Gmbh, Elisabethinen, Linz
  - Uniklinikum Salzburg (LKH) Universitatsklinik fur Innere Medizin III, Salzburg
  - Medical University of Vienna, Vienna
  - Hanusch Krankenhaus, Vienna
- Belgium (5):
  - AZ St.-Elisabeth Herentals vzw, Herentals, Antwerp
  - Hopital De Jolimont, Haine-Saint-Paul, Hainaut
  - Universitair Ziekenhuis (UZ) Gent/ Ghent University Hospital, Ghent, Oost-Vlaanderen
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Institut Jules Bordet, Brussels
- Brazil (17):
  - Ensino e Terapia de Inovacao Clinica Amo (Etica), Salvador, Estado de Bahia
  - Instituto Mario Pena de Ensino Pesquisa e Inovacao, Belo Horizonte, Minas Gerais
  - Liga Norte Riograndense Contra o Cancer, Natal, Rio Grande do Norte
  - Instituto do Cancer em Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Hematologia e Oncologia, Joinville, Santa Catarina
  - Animi Unidade de Tratamento Oncologico Ltda, Lages, Santa Catarina
  - Fundacao Pio XII Hospital de Amor, Barretos, São Paulo
  - Amaral Carvalho Hospital, Jaú, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto da Universidade de Sao Paulo, Ribeirão Preto, São Paulo
  - Instituto DOr de Pesquisa e Ensino Df Star, Brasília
  - Instituto Nacional de Cancer Jose Alencar Gomes da Silva, Rio de Janeiro
  - Instituto Americas, Rio de Janeiro
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - AC Camargo Cancer Center, São Paulo
  - Clinical Hospital of Medicine School at Sao Paulo University, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo
- Canada (5):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Cisss de la Monteregie-Centre, Greenfield Park, Quebec
  - CHU de Quebec - Universite Laval, Québec, Quebec
  - Ciusss de Lestrie - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
- Chile (4):
  - Fundacion Arturo Lopez Perez, Santiago, Santiago Metropolitan
  - Inmunocel, Santiago, Santiago Metropolitan
  - Clinica Alemana de Santiago, Santiago, Santiago Metropolitan
  - Centro Oncologia de Precision Universidad Mayor, Santiago
- Czechia (3):
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Kralovske Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice, Prague
- France (12):
  - Centre Hospitalier Universitaire (CHU) Rennes, Rennes, Brittany Region
  - Centre Hospitalier Regional Universitaire de Tours, Tours, Centre-Val de Loire
  - Nantes University Hospital, Nantes, Pays de la Loire Region
  - Hopital de la Conception, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Universitaire Angers, Angers
  - Institut Paoli Calmettes, Marseille
  - Hopital Saint Louis, Paris
  - Hopital Saint-Antoine, Paris
  - Centre Hospitalier Universitaire (CHU) de Poitiers, Poitiers
  - Institut de Cancerologie Strasbourg Europe (ICANS), Strasbourg
  - Hopital Victor Dupouy Argenteuil, Argenteuil, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region
- Germany (9):
  - Robert-Bosch-Krankenhaus, Stuttgart, Baden-Wurttemberg
  - University Hospital Wurzburg, Würzburg, Bavaria
  - Kliniken Ostalb Stauferklinikum Schwab Gmund, Mutlangen, Gmund
  - Clinic Frankfurt (Oder), Frankfurt am Main, Hesse
  - Universitatsmedizin der Johannes-Gutenberg Universitat Mainz, Mainz, Rhineland-Palatinate
  - Hematological Praxis Dresden, Dresden, Saxony
  - Charite Universitatsmedizin Berlin Campus Benjamin Franklin, Berlin
  - University Hospital Carl Gustav Carus, Dresden
  - Stadtisches Krankenhaus Kiel, Kiel
- Israel (7):
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Bnai Zion Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - Istituto Romagnolo Per Lo Studio Dei Tumori, Meldola, Forli Cesena
  - Irccs Aou Di Bologna- Policlinico Di Sant'Orsola Malpighi, Bologna, Italia
  - Pia Fondazione Panico, Tricase, Lecce
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - Candiolo Cancer Institute, FPO, IRCCS, Candiolo, Torino
  - UOC Ematologia e Terapia Cellulare - PO Mazzoni AST Ascoli Piceno, Ascoli Piceno
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Istituto Europeo di Oncologia, Milan
  - Federico II University, Napoli
  - AOU Maggiore della Carita-SCDU Ematologia, Novara
  - UO Ematologia Ravenna, Ravenna
  - Santa Maria della Misericordia, Udine
  - Ospedale dell'Angelo - Varese, Varese
- Poland (10):
  - Specjalistyczny Szpital im A. Sokolowskiego w Walbrzychu, Wałbrzych, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny, Wroclaw, Lower Silesian Voivodeship
  - Pratia MCM Krakow, Krakow, Malopolska
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Aidport, Skorzewo, Wielkopolska
  - Cm Pratia Poznan, Skorzewo, Wielkopolska
  - Pratia Onkologia Katowice, Katowice
  - Copernicus Memorial Hospital, Lodz
  - Centrum Innowacyjnych Terapii Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy Warszawa, Warsaw
- South Korea (7):
  - Center for Hematologic Malignancy, Goyang-si, Gyeonggi-do
  - St. Vincents Hospital - The Catholic University of Korea, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Jeonbuk National University Hospital, Jeonju
  - Seoul St. Mary's Hospital, Seoul
- Spain (27):
  - University Hospital of Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitario Virgen De La Victoria Malaga, Málaga, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Son Espases University Hospital, Palma, Balearic Islands
  - Cruces University Hospital (Hospital Universitario Cruces), Barakaldo, Bizkaia
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Universitario de a Coruna, A Coruña, Galicia
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Clinico Universitario Virgen De La Arrixaca, El Palmar, Murcia
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central De Asturias, Oviedo, Principality of Asturias
  - University Hospital Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Virgen De Las Nieves De Granada, Granada
  - Gregorio Maranon, Madrid
  - Clinica Universidad de Navarra, Madrid
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - University Hospital & Research Institute, Madrid
  - Hospital Universitario HM Sanchinarro, Servicio de Hematologia, Madrid
  - Morales Meseguer Hospital, Murcia
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario de Salamanca, Salamanca
  - University Hospital Virgen del Rocio, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Clinico Universitario Valencia, Valencia
  - Hospital Universitari and Politecnic La Fe, Valencia
  - Hospital Clinico Lozano Blesa, Zaragoza
- Switzerland (5):
  - Kantonsspital Baden, Baden, Canton of Aargau
  - Cantonal Hospital St Gallen, Sankt Gallen, Canton of St. Gallen
  - Kantonsspital Winterthur Medical Oncology, Winterthur, Schweiz
  - University Hospital Basel, Basel
  - Inselspital Bern University Hospital, Bern
- Taiwan (12):
  - Chang Gung Medical Foundation Chia Yi Branch, Buzi, Chiayi County
  - Chang Gung Memorial Hospital Linkou, Taoyuan, Guishan District
  - Changhua Christian Hospital, Changhua
  - Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - Taichung General Veterans Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
- Turkey (Türkiye) (13):
  - Ankara University Faculty of Medicine, Mamak, Ankara
  - Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Yenimahalle, Ankara
  - Gazi University, Ankara, Central Anatolia
  - VM Medical Park Mersin Hospital, Mezitli, Mersin
  - Tekirdag Namik Kemal University Hospital, Tekirdağ, Suleymanpasa
  - Liv Hospital Ankara, Ankara
  - VKV American Hopital, Istanbul
  - Istanbul University Istanbul Faculty of Medicine, Istanbul
  - Ege University, Izmir
  - Erci̇yes Uni̇versi̇ty, Kayseri
  - Sakarya University Medical Faculty, Sakarya
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
  - Zonguldak Bulent Ecevit University, Zonguldak
- United Kingdom (6):
  - Royal Cornwall Hospital NHS Trust, Truro, Cornwall
  - Derriford Hospital and the Royal Eye Infirmary, Plymouth, Devon
  - University Hospitals Dorset, Bournemouth, Dorset
  - Beatson West of Scotland Cancer Centre, Glasgow, Lanarkshire
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Barking, Havering and Redbridge University Hospitals NHS Trust, Romford

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: OLYMPIA — https://olympiastudies.com/en-us